CLINICAL TRIAL: NCT07250269
Title: A Phase 1b Study of GC012F, a Chimeric Antigen Receptor T Cell Therapy Targeting CD19 and B-cell Maturation Antigen in Chinese Participants With Relapsed or Refractory AL Amyloidosis
Brief Title: Study of GC012F, CAR-T Therapy Targeting CD19 and BCMA in Chinese Participants With Relapsed or Refractory AL Amyloidosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Collaborators: Suzhou Gracell Biotechnologies Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D831AC00002
Record Dates: First submitted 2025-10-21; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC012F (Experimental): GC012F Injection
  Interventions: Drug: GC012F Injection

INTERVENTIONS:
Drug: GC012F Injection — The investigational agent, GC012F, is an autologous BCMA/CD19 dual directed CAR product under investigation for the treatment of patients with RRMM, ELMM, SLE, and B NHL.
  Other Names: AZD0120

SUMMARY:
This is a Phase 1b open-label, multicenter, non-randomized study of GC012F, a CD19/BCMA dual CAR T cell therapy, in adult participants with relapsed/refractory AL amyloidosis.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multicenter, non-randomized study to evaluate the safety, tolerability, and efficacy of GC012F in adult participants with relapsed/refractory AL amyloidosis. A single-arm design was chosen for the study due to the absence of approved therapies for use as a concurrent control for this patient population. In the study, the safety of different doses of GC012F will be evaluated and the RP2D will be selected based on the totality of clinical safety, preliminary efficacy, CK and PD data.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed histopathological diagnosis of AL amyloidosis
2. One or more organs currently or historically impacted by AL amyloidosis according to consensus guidelines
3. Measurable hematologic disease: dFLC > 20 mg/L or serum M-protein > 5g/L
4. Relapsed disease or refractory disease defined as a need for additional therapy after at least 1 line of anti-plasma cell-directed therapy.
5. ECOG performance status of 0 to 1
6. Must be able and willing to adhere to the study visit schedule and other protocol requirements
7. Women of child-bearing potential (WCBP) must have a negative serum pregnancy test prior to treatment. All sexually active WCBP and all sexually active male subjects must agree to use effective methods of birth control throughout the study.

Exclusion Criteria:

1. Have any other form of amyloidosis other than AL amyloidosis
2. Mayo Stage IIIb AL amyloidosis
3. Oxygen saturation < 95% on room air
4. Systolic blood pressure <100mmHg
5. Cardiac exclusion criteria:

   1. Mayo Stage IIIb AL amyloidosis (Wechalekar, 2013)
   2. NT-proBNP levels as follows:

NT-proBNP ≥ 2000 ng/L (for dose escalation portion) NT-proBNP < 2000 and > 5000 ng/L (for dose extension portion) c. High-sensitivity cardiac troponin T > 75 ng/L d. NYHA class III or IV 5. Extensive GI involvement with evidence of active GI bleeding/risk of bleeding as determined by Investigator 6. Prior therapies:

1. CAR T cell therapy directed at any target
2. Prior BCMA-targeting therapy
3. Prior treatment with any approved or investigational T cell engaging therapies (including T cell-directed bispecific or trispecific therapies) at any target within the last 6 months.

7. Toxicity from previous anti-cancer or anti-PC-directed therapy did not resolve to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy.

8. Active plasma cell leukemia at the time of screening 9. Multiple myeloma defined as clonal bone marrow PCs ≥10% and any one or more of the following myeloma defining events (deemed as attributable to multiple myeloma by Investigator) (Rajkumar, 2014) 10. Seropositive for HIV 11. Serologic status reflecting active hepatitis B or C:

1. Positive HBsAg, or
2. Patients with positive core antibody (anti-HBc) and HBV-DNA positive.
3. Patients with positive hepatitis C antibody and HCV RNA positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2028-11-24 (Estimated); Study Completion 2028-11-24 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With incidence and severity of Treatment-emergent Adverse Events | Through study completion, an average of 2 years
Proportion of Participants Experiencing a Complete Response | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Levels of AZD0120 in blood over time in participants with AL amyloidosis | Through study completion, an average of 2 years
Percentage of participants achieving hematologic response | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Suzhou
  - Research Site, Wenzhou
  - Research Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/